CLINICAL TRIAL: NCT01762358
Title: Effectiveness of a Non-invasive Therapy for Treating Fully Ruptured Anterior Cruciate Ligaments in the Knee by Using MRI, Functional Tests and Scores: A Randomized Controlled Trial
Brief Title: Khalifa Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Andreas Sandner-Kiesling , MD, Univ.Prof.Dr., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KhalMUG1
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Total Rupture of the Anterior Cruciate Ligament in the Knee
Keywords: ACL; Ligament; Knee
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Therapy (Active Comparator): Standardized physiotherapy for 12 times (15 patients)
  Interventions: Other: Physiotherapy
- Standard + Khalifa (Experimental): Initial one hour Khalifa therapy followed by twelve times standardized Physiotherapy (15 patients)
  Interventions: Other: Khalifa's therapy

INTERVENTIONS:
Other: Khalifa's therapy — One hour of Khalifa's therapy which is specially applied pressure to the skin
  Arms: Standard + Khalifa
Other: Physiotherapy — Twelve times standardized Physiotherapy
  Arms: Standard Therapy

SUMMARY:
The primary hypothesis is that Khalifa's therapy brings additional benefit compared to standard therapy (physiotherapy) for patients with a ruptured anterior cruciate ligament (ACL).

DETAILED DESCRIPTION:
Mohamed Khalifa, a therapist from Hallein (Austria), has been working since 30 years with a self-developed manual technique for treating injuries of the musculoskeletal system especially of the knee by applying high pressure to the skin in the area of the injury. This pressure is applied in various amplitudes and frequencies.

International top athletes from various disciplines reported a rapid pain relief, and even full recovery, immediately after his one hour treatment.

Prior to the investigators' study, the investigators evaluated one pilot patient with a complete ACL rupture after a soccer game with Magnet-Resonance-Imaging (MRI) and clinical tests. This patient was physically immobile and reported pain especially when stretching and bending the knee. After one hour of treatment from Khalifa the signs of the injury like the stretching / bending inhibition and pain were gone immediately. Three months after the treatment, an evaluation of the knee with MRI showed an end-to-end continuous ACL with homogeneous signal and the clinical tests confirmed the stability of the knee.

With this study the investigators will evaluate the possibility of influencing the healing of a completely ruptured ACL of the knee by one single special local pressure treatment to the skin for 60 min.

ELIGIBILITY:
Inclusion Criteria:

* totally ruptured ACL - MRI verified, 4 weeks old as a maximum
* knee function: Any functional inhibition (stretching, bending or load)
* BMI: 18-28
* athletically active

Exclusion Criteria:

* any surgical procedures at the injured knee at any previous time
* any acute surgical indication
* diabetes mellitus and/or high blood pressure
* any permanent drug treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
ACL Morphology | 3 months after 1st therapy
  Magnet resonance images: end-to-end homogeneous anterior cruciate ligament
Knee function | 24 hours and 3 months after 1st therapy
  IKDC-Score (International Knee Documentation Comite) clinical / physical examination KT-1000 evaluation

SECONDARY OUTCOMES:
Life Quality | 24 hours, 3 months
  A Visual Analogue Scale was used to evaluate: Pain and Well-being

OTHER OUTCOMES:
Confidence | 24 hours, 3 months
  Confidence in therapists / doctors were evaluated by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Engelbert Wallenböck, MD, Principal Investigator — UKH Graz; Robert Pehn, MD, Principal Investigator — AKH Kirchdorf; Frank Schneider, MD, Principal Investigator — LKH Graz; Andreas Kastner, MD, Principal Investigator — AKH Linz; Andreas Sandner, MD, Study Director — Med Uni Graz
Locations (4):
- Austria (4):
  - LKH, Graz
  - UKH, Graz
  - LKH, Kirchdorf
  - AKH, Linz